CLINICAL TRIAL: NCT07296692
Title: Effect of a Nutritional Formula Composed of Proteins and Carbohydrates on Gastric Emptying in Elderly Individuals: a Randomized, Crossover, Triple-blind Clinical Trial.
Brief Title: Effect of a Nutritional Formula Composed of Proteins and Carbohydrates on Gastric Emptying in Elderly Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Nestle Health Science (Industry)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, Phd, Federal University of Minas Gerais
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 91081525.0.0000.5149
Record Dates: First submitted 2025-09-26; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Gastric Emptying
Keywords: proteíns; elderly; gastric emptying; scintigraphy
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formula (Experimental): In this arm, participants will undergo scintigraphy after consuming the formula composed of carbohydrates and proteins, over a period of 3 hours (immediately after ingestion and 1 to 3 hours post-ingestion). After the first arm, a 7-day washout period will be implemented
  Interventions: Dietary Supplement: Nutren Fresh
- Placebo (Placebo Comparator): In this arm, participants will undergo scintigraphy after consuming the formula composed only of carbohydrates, over a period of 3 hours (immediately after ingestion and 1 to 3 hours post-ingestion). After the first arm, a 7-day washout period will be implemented.
  Interventions: Dietary Supplement: Maltodextrin (Placebo)

INTERVENTIONS:
Dietary Supplement: Nutren Fresh — In this intervention, participants will receive 200 ml of the nutritional formula.
  Arms: Formula
Dietary Supplement: Maltodextrin (Placebo) — In this intervention, participants will receive 200 ml of maltodextrin.
  Arms: Placebo

SUMMARY:
The objective of this clinical trial is to evaluate the effect of a nutritional formula composed of carbohydrates and proteins on gastric emptying in elderly individuals aged between 60 and 90 years. The main questions this study aims to answer are:

* Does the nutritional formula composed of carbohydrates and proteins delay gastric emptying when compared to a formula composed only of carbohydrates?
* Does the formula composed of carbohydrates and proteins cause gastrointestinal symptoms in the study population?

The researchers will compare both formulas (carbohydrates and proteins vs. carbohydrates only) to answer the main question.

Participants will be required to:

* Attend the Nuclear Medicine Department after an 8-hour fast, on two separate days with a minimum interval of seven days for scintigraphy procedures.
* Consume the offered formula in a randomized and blinded manner.
* Report any gastrointestinal symptoms and complete visual analog scales for sensations such as hunger, satiety, and desire to eat.

DETAILED DESCRIPTION:
Preoperative fasting (POF) is defined as the absence of food or fluid intake in the hours preceding surgery. POF is recommended to minimize the risk of aspiration of gastric contents and related complications. However, the incidence of such complications is low. Prolonged fasting can have adverse effects on the patient's health, such as headache, dehydration, hypovolemia, and hypoglycemia, potentially compromising postoperative recovery.

Shortening the fasting period with nutrient-containing clear liquids administered up to two hours before surgery has been shown to be a safe and beneficial alternative. Additionally, the use of formulas containing not only carbohydrates but also proteins has been tested in order to promote further benefits, such as attenuation of negative nitrogen balance and improvement in patient prognosis.

Given the increasing life expectancy of the population, the number of surgeries in elderly patients is also growing. This is coupled with the fact that aging is associated with physiological reductions in gastric emptying rate and hydrochloric acid secretion, requiring greater care in determining appropriate POF duration.

In this context, the objective of this study is to compare the gastric emptying (GE) of elderly volunteers after consuming a standard formula containing only carbohydrates with another formula composed of both carbohydrates and proteins, administered at two different time points.

This is a randomized, crossover, triple-blind clinical trial involving elderly individuals. The study will include individuals aged 60 years or older, who are non-smokers and have no prior diagnosis of conditions that affect gastric emptying. Patients will be randomized into group A or B to determine the order of interventions. Each volunteer will receive the designated formula in a randomized and blinded manner on the study day, with the formula containing approximately 1 mCi of 99mTc-sodium phytate.

Immediately after finishing the formula intake, participants will undergo the first scintigraphic imaging (T0). Additional scintigraphic images will be taken at 60, 120, and 180 minutes post-ingestion. The mean time to empty half of the gastric content will be assessed, with values less than 25 minutes considered normal.

Gastrointestinal symptoms, as well as sensations of hunger, satiety, and desire to eat, will also be assessed using visual analog scales (VAS), applied on study days. Capillary blood glucose will be measured using a portable glucometer.

Data will be analyzed using statistical software, and normality will be tested to determine the appropriate statistical tests. P-values ≥ 0.05 will be considered statistically significant.

The sample size will be calculated based on a pilot study involving at least 25 volunteers, since there are no similar prior studies. The parameters from this pilot study may then be used to determine the final sample size.

ELIGIBILITY:
Inclusion Criteria:

* Elderly individuals aged between 60 and 90 years
* Non-smokers
* No prior diagnosis of conditions that affect gastric emptying, such as:
* Gastroesophageal reflux
* Gastroparesis
* Untreated Helicobacter pylori (H. pylori) infection
* Stomach cancer
* Esophageal cancer

Exclusion Criteria:

* Volunteers who do not meet the inclusion criteria
* Refusal to sign the informed consent form (ICF)
* Volunteers with obesity (BMI over 35 kg/m²)
* Volunteers who do not eat orally or have a prior diagnosis of delayed gastric emptying and are on routine use of prokinetic medications
* Individuals diagnosed with Alzheimer's or Parkinson's disease

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Gastric Emptying | On day 1 and day 2 of the protocol.
  Gastric emptying will be assessed through scintigraphic imaging obtained immediately after formula consumption and every hour for three hours.

SECONDARY OUTCOMES:
Gastrointestinal symptoms and sensations of hungry, saciety and desire to eat | Immediately after formula ingestion, and at 60, 120, and 180 minutes post-ingestion.
  Use of numerical visual analog scales (from 0 to 10, with 0 indicating no symptoms and 10 indicating severe symptoms.), where the volunteer will indicate the presence and intensity of gastrointestinal symptoms (heartburn, nausea, burning sensation, etc.) and sensations of hunger, satiety, and desire to eat.
Blood glucose | This assessment will be conducted with the patient in a fasting state, immediately after formula ingestion, and at 60, 120, and 180 minutes post-ingestion on each protocol day.
  To assess capillary blood glucose using a portable glucometer.

CONTACTS AND LOCATIONS:
Overall Officials: Simone de Vasconcelos Generoso Generoso, Phd, Principal Investigator — Department of Nutrition, Federal University of Minas Gerais
Locations (1):
- School of Nursing, Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No